CLINICAL TRIAL: NCT04350814
Title: Efficacy of a Self-Compassion Intervention to Prevent Relapse and Recurrence of Depression: Fostering Trait Resilience to Disrupt the Cycle of Depression
Brief Title: The Self-Compassion Online - Preventing Depression Trial
Acronym: SCOPE
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Regina (Other)
Collaborators: Saskatchewan Health Research Foundation (Other); University of Amsterdam (Other); University of Oxford (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Prevention
Other Study IDs: 2018-229
Record Dates: First submitted 2020-04-14; First posted 2020-04-17 (Actual); Last update posted 2024-05-08 (Actual); Status verified 2024-05

CONDITIONS: Depression
MeSH Terms: conditions — Depression

STUDY DESIGN:
Intervention Model Description: The investigators will randomly assign participants to one of two conditions, and monitor their symptoms for 12 months. After the 12-months assessment period is complete, the investigators will offer the intervention to participants assigned to the active control condition to use at their own discretion.
Who Masked: Investigator
Masking Description: No research assistants involved in participant assessment, nor is the primary investigator, aware of which condition participants are assigned to. This masking will be monitored and conducted by a lab staff member not directly involved in the study.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Self-Compassion Intervention Arm (Experimental): Participants randomized to this condition will receive access to the audio Mindful Self-Compassion self-help intervention. The intervention is 7 weeks in duration (with a pacing of one lesson per week) and participants are asked to complete study measures once each week of the intervention.
  Interventions: Behavioral: Self-Compassion Step by Step
- Self-Reflection (Active Comparator): Participants randomized to this active control condition will be asked to complete study measures at the same assessment intervals as those in the experimental arm. In addition to completing the measures, participants in the Self-Reflection Active Control condition will be asked to reflect on their self-reported symptoms and changes they may have experienced between assessment intervals.
  Interventions: Behavioral: Self-Reflection Active Control

INTERVENTIONS:
Behavioral: Self-Compassion Step by Step — This is a 6-lesson self-guided audio program by Dr. Kristen Neff (2013)
  Arms: Self-Compassion Intervention Arm
Behavioral: Self-Reflection Active Control — Participants randomized to this active control condition will be asked to complete study measures at the same intervals as those assigned to the intervention condition. In addition to completing study questionnaires, participants in this arm will also be invited to reflect on their weekly reported symptoms, whether they experienced changed, what they believe these changes are attributed to, etc.
  Arms: Self-Reflection

SUMMARY:
Purpose: Depression affects 12.6% of Canadians at some point in their life. Depression is associated with staggering personal and economic costs. There are several treatments that have been shown to treat episodes of depression when they occur. Unfortunately, more than half who respond to these treatments go on to re-experience an episode of depression. Even with psychological and pharmacological interventions designed to prevent future episodes, relapse and recurrence of the disorder remain alarmingly high. A patient-focused and self-directed intervention that harnesses the effects of an Eastern-influenced concept, called self-compassion, has shown tremendous promise in treating acute depression. Self-compassion is being moved by one's own suffering, and a desire to alleviate such suffering.

Objectives: In the proposed project, the investigators will examine whether a self-compassion intervention is effective in preventing relapse/recurrence of depression over a 12-month period among people who are at high risk for relapse. The investigators will also examine whether the intervention works to prevent depression by increasing the innate ability to bounce back from stress, a concept known as resilience.

Methodology: 120 participants with a history of depression will be randomly assigned to the self-compassion intervention or a self-assessment reflection condition, and their respective relapse rates will be examined over a period of 12 months.

Importance to Research: This will be the first study to examine the effects of self-compassion as a preventive intervention for depression.

Impact on health: If successful, this new intervention can be used by thousands of people in Saskatchewan and Canada who are at risk for depression relapse.

ELIGIBILITY:
Inclusion Criteria:

* To be eligible to participate in the study, participants must be: a) 18 years old or older; b) have experienced at least one episode of depression; and c) exhibit elevated residual symptoms of depression-as indicated by a score of 5 or more on the Patient Health Questionnaire-9 (PHQ-9; Kroenke, Spitzer, & Williams, 2001). As the majority of people experience both depression and anxiety symptoms concurrently, participants experiencing elevated anxiety symptoms will not be excluded from the study.

Exclusion Criteria:

* Participants will be excluded from the study if they indicate: a) a current diagnosis MDD, substance use disorder, psychosis, or mania in accordance with the Diagnostic and Statistical Manual of Mental Disorders-5 (DSM-5; American Psychiatric Association, 2013); b) the presence of major health conditions (e.g., cardiovascular diseases, cancer, hypothyroidism, etc.); and c) currently undergoing psychological or pharmacological treatment at the time of recruitment

Ages: 18 Years to 79 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 158 (Actual)
Dates: Start 2020-03-01 (Actual); Primary Completion 2023-12-01 (Actual); Study Completion 2024-05-01 (Actual)

PRIMARY OUTCOMES:
Longitudinal Interval Follow-UP Evaluation - Structured Clinical Interview (LIFE-SCID) | 12 Months
  Proportional rates of individuals meeting criteria for major depression episode in accordance with the LIFE-SCID post randomization over 12-months across two conditions.
  This measure is a diagnostic interview: Outcomes are binary (diagnosis vs. no diagnosis)
Weeks to Relapse | 12 Months
  Time in weeks to confirmed MDE relapse during the assessment period
  This is a linear calculation of how many weeks participants stayed diagnosis free (higher is more weeks without a depressive relapse/recurrence).
Scores on the Patient Health Questionnaire - 9 over 12-months | 12 Months
  Differences in depressive symptoms among those randomized to the intervention or active control condition at the 12-month assessment period
  This measure is a diagnostic interview: Outcomes are binary (diagnosis vs. no diagnosis)

SECONDARY OUTCOMES:
Self-Compassion Scale (SCS) | Post-intervention, 3, 6, 9, and 12 Months
  This is a measure of dispositional self-compassion. Scores range from 12-60, with higher scores indicative of greater dispositional self-compassion.
Five-Facet Mindfulness Questionnaire-15 | Post-intervention, 3, 6, 9, and 12 Months
  This is a measure of dispositional mindfulness skills. Scores range from 15-75, with higher scores indicative of greater dispositional mindfulness.
Experiences Questionnaire-Decentering | Post-intervention, 3, 6, 9, and 12 Months
  This is a measure of dispositional decentring abilities (viewing all experiences, including internal experiences, as passing events). Scores range from 12-48, with higher scores indicative of greater decentring.
Fears of Compassion Scales (FCS) | Post-intervention, 3, 6, 9, and 12 Months
  This is a measure of the fear of showing one's self compassion. Scores range from 10 to 50, with higher scores indicative of greater fears of self compassion.

CONTACTS AND LOCATIONS:
Overall Officials: Shadi Beshai, PhD, Principal Investigator — University of Regina
Locations (2):
- Canada (2):
  - University of Regina, Regina, Saskatchewan
  - DCC Lab, Regina

IPD SHARING:
Plan to Share IPD: No